CLINICAL TRIAL: NCT00586963
Title: How Does Proton Pump Inhibitor Therapy Impact Quality of Life in Patients Newly Diagnosed With Erosive Reflux Esophagitis?
Brief Title: Proton Pump Inhibitor (PPI) Therapy for Newly Diagnosed Esophagitis
Acronym: EE
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Yvonne Romero, Mayo Clinic
Other Study IDs: 07-006142; IRUSESOM0488
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Erosive Esophagitis; Reflux Esophagitis; GERD
Keywords: Erosive Esophagitis; Reflux Esophagitis; GERD
MeSH Terms: conditions — Esophagitis, Peptic; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is being done to for two reasons:

* To learn about the effects (good and bad) esomeprazole (an FDA approved drug for reflux esophagitis) has on your esophagus when taken correctly.
* To learn about the quality of life changes (good and bad) you may experience with this medication.

DETAILED DESCRIPTION:
The plan is to have 50 people take part in this study at Mayo Clinic Rochester. This research study is looking at people who have a new condition called erosive reflux esophagitis. Esophagitis is defined as mucosal damage produced by the abnormal reflux of gastric contents into the esophagus. Acid reflux, over time, can wear away or erode the lining of your esophagus. This condition is called erosive esophagitis. The treating physician may start you on prescription strength acid reducing group of medications called Proton Pump Inhibitors (PPI). PPI medications can provide 24-hour relief from your painful heartburn symptoms and it can help you heal the erosions in the esophagus that acid reflux may cause.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Have either mild-to-moderate erosive reflux esophagitis
* Meet criteria for GERD symptoms.

Exclusion Criteria:

* Patients already on esomeprazole therapy, have previously failed to respond to esomeprazole, or are intolerant to PPI therapy.
* Patients expected to travel outside of the United States during the initial 8 weeks of PPI therapy.
* Pregnant women will be excluded as PPI's are not thought safe for the fetus (Pregnancy Category C). - Children younger than 18 years of age will be excluded.
* Other vulnerable populations, such as those with diminished mental acuity, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients age 18 and older, diagnosed with reflux esophagitis, being seen at Mayo Clinic Rocheser.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Romero, MD., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States